CLINICAL TRIAL: NCT02717754
Title: A Multiple-Center, Randomized, Double-blind, Multiple-Dose, Placebo-Controlled, Parallel-Group Study to Investigate the Safety, Tolerability, and Pharmacokinetics of RO0640796 (Oseltamivir) and Its Carboxylate Metabolite, RO0640802, Following Intravenous Administrations in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics (PK) of Oseltamivir and Its Carboxylate Metabolite, RO0640802 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NP25140
Record Dates: First submitted 2016-03-20; First posted 2016-03-24 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Oseltamivir 100 mg (Experimental): Participants will receive 100 mg oseltamivir intravenous BID for 5 days.
  Interventions: Drug: Oseltamivir
- Oseltamivir 200 mg (Experimental): Participants will receive 200 mg oseltamivir intravenous BID for 5 days.
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator): Participants will receive oseltamivir matched placebo intravenous BID for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir will be administered at 100 or 200 mg intravenous BID for 5 days.
  Other Names: Tamiflu, RO0640796
  Arms: Oseltamivir 100 mg; Oseltamivir 200 mg
Drug: Placebo — Oseltamivir matched placebo will be administered intravenous for 5 days.
  Arms: Placebo

SUMMARY:
This multi-center, randomized, double-blind, multiple-dose, placebo-controlled, parallel-group study will assess the safety and PK of oseltamivir (Tamiflu) and its carboxylate metabolite, RO0640802 in healthy participants. Participants will be randomized to receive 100 milligrams (mg) oseltamivir, 200 mg oseltamivir, or placebo, all administered intravenously twice daily (BID). The anticipated time on study treatment is 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Body Mass Index (BMI) 18-34 kilograms per meter square (kg/m^2), inclusive
* Male participants who are willing to use barrier contraception for the duration of the study and for 3 months following the end of treatment
* Female participants who are of non-child bearing potential
* Female participants who are of child bearing potential utilizing two effective methods of contraception for the duration of the study and for 3 months following the end of treatment

Exclusion Criteria:

* Evidence of clinically significant disease or disorder (for example, renal, cardiac, bronchopulmonary)
* Any other condition or disease which would place the participant at undue risk, or interfere with the assessment, or with the ability of the participant to complete the study
* Clinically significant orthostatic hypotension present at screening or history of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or lightheadedness.
* Participants with abnormal electrocardiogram (ECG), bradycardia or mean QTc at screening
* Positive result for Hepatitis B, Hepatitis C, human immunodeficiency virus (HIV) 1 or 2 at screening
* Renal impairment
* Transplant recipients
* A known clinically relevant history of allergy or hypersensitivity
* Any clinically relevant abnormal laboratory test results
* A clinically relevant history of abuse of alcohol or other drugs of abuse
* Any major illness within 30 days prior to the screening examination
* Smoking of more than 10 cigarettes a day or an equivalent amount of tobacco in the form of cigars or pipe
* Participation in a clinical study with an investigational drug within 3 months prior to Day 1
* Donation/loss of more than 500 milliliters (mL) of blood within 3 months prior to Day 1
* Positive pregnancy test at screening or Day -1 and lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Little Rock, Arkansas
  - Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 99 participants were included in study, but as first 50 participants were administered infusion incorrectly thus only 49 participants were considered evaluable for pharmacokinetics. The 50 participants were reported for safety under arm groups placebo (incorrect infusion duration), oseltamivir 100 or 200 mg (incorrect infusion duration).
Groups:
- Placebo: Participants received oseltamivir matched placebo twice daily (BID) for 5 days.
- Oseltamivir 100 mg: Participants received 100 milligrams (mg) oseltamivir intravenous BID for 5 days.
- Oseltamivir 200 mg: Participants received 200 mg oseltamivir intravenous BID for 5 days.
- Placebo (Incorrect Infusion Duration): Participants were randomized to receive oseltamivir matched placebo intravenous BID for 5 days but received incorrect infusion duration.
- Oseltamivir 100 mg (Incorrect Infusion Duration): Participants were randomized to receive oseltamivir 100 mg intravenous BID for 5 days but received incorrect infusion duration.
- Oseltamivir 200 mg (Incorrect Infusion Duration): Participants were randomized to receive oseltamivir 200 mg intravenous BID for 5 days but received incorrect infusion duration.
Period: Overall Study
Arm/Group | Placebo | Oseltamivir 100 mg | Oseltamivir 200 mg | Placebo (Incorrect Infusion Duration) | Oseltamivir 100 mg (Incorrect Infusion Duration) | Oseltamivir 200 mg (Incorrect Infusion Duration)
Started | 10 | 19 | 20 | 10 | 20 | 20
Completed | 10 | 19 | 20 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 10 | 20 | 20
Not completed — Incorrect Infusion Duration | 0 | 0 | 0 | 10 | 20 | 20

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug and have a safety assessment performed after initiation of treatment.
Groups:
- Placebo: Participants received oseltamivir matched placebo BID for 5 days.
- Oseltamivir 100 mg: Participants received 100 mg oseltamivir intravenous BID for 5 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Oseltamivir 100 mg | Oseltamivir 200 mg | Placebo (Incorrect Infusion Duration) | Oseltamivir 100 mg (Incorrect Infusion Duration) | Oseltamivir 200 mg (Incorrect Infusion Duration) | Total
Number analyzed (Participants) | 10 | 19 | 20 | 10 | 20 | 20 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.19) | 28.3 (6.97) | 30.2 (7.73) | 29.7 (7.90) | 31.1 (7.80) | 28.6 (8.09) | 29.4040 (7.44904)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 4 | 1 | 3 | 4 | 27
  Male | 5 | 9 | 16 | 9 | 17 | 16 | 72

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 12 Hour (AUC0-12h) of Oseltamivir and RO0640802 at Steady State
Description: AUC is a measure of the plasma concentration of the drug over time. AUC is presented in nanogram times (*) hour per milliliter (ng*hour/mL). RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 5
Population: Pharmacokinetic (PK) analysis population included all participants who were dosed correctly. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng*hour/mL
  Oseltamivir | 581 (178) | 1143 (178)
  RO0640802 | 4147 (742) | 7966 (1427)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Oseltamivir and RO0640802 at Steady State
Description: Cmax is the maximum observed plasma concentration, presented in nanogram per milliliter (ng/mL). RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng/mL
  Oseltamivir | 266 (73.1) | 496 (69.7)
  RO0640802 | 488 (84.1) | 960 (178)

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Oseltamivir and RO0640802
Description: AUC is a measure of the plasma concentration of the drug over time. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng*hour/mL
  Oseltamivir | 612 (134) | 1139 (220)
  RO0640802 | 3606 (761) | 7336 (1952)

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of Oseltamivir and RO0640802
Description: as for outcome 3
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1 and Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng*hour/mL
  Day 1: Oseltamivir | 609 (134) | 1136 (220)
  Day 1: RO0640802 | 2273 (405) | 4566 (714)
  Day 5: Oseltamivir | 580 (178) | 1142 (178)
  Day 5: RO0640802 | 4127 (738) | 7932 (1417)

5. Secondary Outcome: Cmax of Oseltamivir and RO0640802
Description: Cmax is the maximum observed plasma concentration. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng/mL
  Oseltamivir | 284 (54.3) | 503 (93.1)
  RO0640802 | 301 (69.8) | 577 (88.9)

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Oseltamivir and RO0640802
Description: Tmax is time of observed maximum plasma concentration. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1 and Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
hour
  Day 1: Oseltamivir | 1.85 (0.377) | 1.65 (0.491)
  Day 1: RO0640802 | 3.90 (0.91) | 3.95 (1.28)
  Day 5: Oseltamivir | 1.64 (0.492) | 1.81 (0.416)
  Day 5: RO0640802 | 3.69 (0.917) | 3.41 (0.851)

7. Secondary Outcome: Half-Life (t1/2) of Oseltamivir and RO0640802
Description: t1/2 is the time measured for the plasma concentration to decrease by one half. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1 and Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
hour
  Day 1: Oseltamivir | 1.22 (0.32) | 1.53 (0.293)
  Day 1: RO0640802 | 6.89 (2.08) | 7.17 (2.19)
  Day 5: Oseltamivir | 1.40 (0.327) | 1.88 (0.457)
  Day 5: RO0640802 | 7.97 (1.82) | 8.17 (2.23)

8. Secondary Outcome: Volume of Distribution (Vd) of Oseltamivir and RO0640802
Description: Vd is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1 and Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
Liter
  Day 1: Oseltamivir | 171 (36.4) | 183 (39)
  Day 1: RO0640802 | 250 (55) | 251 (45.7)
  Day 5: Oseltamivir | 189 (103) | 192 (31.0)
  Day 5: RO0640802 | 266 (58.9) | 280 (65.9)

9. Secondary Outcome: Clearance (CL) of Oseltamivir and RO0640802
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: Predose (0 hour), 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12 hours post dose on Day 1 and Day 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
Liters/hour
  Day 1: Oseltamivir | 289 (55) | 393 (67)
  Day 1: RO0640802 | 26.0 (5.4) | 25.4 (6.1)
  Day 5: Oseltamivir | 192 (74.6) | 179 (30.3)
  Day 5: RO0640802 | 21.7 (3.80) | 22.6 (3.9)

10. Secondary Outcome: Minimum Plasma Concentration (Cmin) of RO0640802
Description: Collection of the 12-hour post-dose sample took place prior to administration of the second daily dose of drug. RO0640802 is the pharmacologically active carboxylate metabolite of oseltamivir.
Time Frame: 12-hour post dose on Day 1, 5 and predose on Day 2, 3, 4, 5
Population: PK analysis population. Only participants who received oseltamivir were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir 100 mg | Oseltamivir 200 mg
Number analyzed (Participants) | 19 | 20
ng/mL
  Day 1 (12-hour post dose) | 131 (29.3) | 264 (59.1)
  Day 2 (Pre dose) | 209 (43.6) | 388 (95.4)
  Day 3 (Pre dose) | 235 (56.3) | 450 (101)
  Day 4 (Pre dose) | 277 (104) | 443 (143)
  Day 5 (Pre dose) | 262 (68.4) | 502 (130.4)
  Day 5 (12-hour post dose) | 238 (61.8) | 458 (110)

ADVERSE EVENTS:
Time Frame: Up to 10 days after last dose of study drug (32 days)
Description: In total 99 participants were included in study, but as first 50 participants were administered infusion incorrectly thus only 49 participants were considered evaluable for pharmacokinetics. The 50 participants were reported for safety under arm groups placebo (incorrect infusion duration), oseltamivir 100 or 200 mg (incorrect infusion duration).
Groups:
- Placebo: Participants received oseltamivir matched placebo for 5 days.
Arm/Group | Placebo | Oseltamivir 100 mg | Oseltamivir 200 mg | Placebo (Incorrect Infusion Duration) | Oseltamivir 100 mg (Incorrect Infusion Duration) | Oseltamivir 200 mg (Incorrect Infusion Duration)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/19 | 0/20 | 0/10 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/10 | 17/19 | 20/20 | 2/10 | 8/20 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Oseltamivir 100 mg (N=19) | Oseltamivir 200 mg (N=20) | Placebo (Incorrect Infusion Duration) (N=10) | Oseltamivir 100 mg (Incorrect Infusion Duration) (N=20) | Oseltamivir 200 mg (Incorrect Infusion Duration) (N=20)
Infusion site pain (General disorders) | 3 | 15 | 15 | 0 | 0 | 1
Infusion site erythema (General disorders) | 1 | 6 | 10 | 0 | 1 | 4
Infusion site swelling (General disorders) | 3 | 3 | 1 | 0 | 0 | 0
Infusion site induration (General disorders) | 0 | 4 | 2 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 2 | 2 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Infusion site anaesthesia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Catheter site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion site coldness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion site warmth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vein disorders (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 9
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 6
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.